CLINICAL TRIAL: NCT04634084
Title: Subacromial Bursa Re-Implantation After Rotator Cuff Repair - A Randomized Controlled Trial
Brief Title: Subacromial Bursa Re-Implantation After Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James M. Gregory, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-1092
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Injuries
Keywords: subacromial bursa
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Procedure: Experimental group(Bursa Implantation)
- Control Group (Active Comparator)
  Interventions: Procedure: Control Group(Standard of Care)

INTERVENTIONS:
Procedure: Experimental group(Bursa Implantation) — Prior to all rotator cuff repairs, a subacromial bursectomy is performed with an oscillating shaver so that the rotator cuff can be visualized and repaired.In the experimental group, instead of being discarded, this minced bursal tissue will be collected via a sterile filtration device attached to the oscillating shaver. The bursal tissue is then placed into a sterile syringe, and reimplanted back onto the bursal surface of the rotator cuff repair at the completion of the case. The arthroscopic fluid is turned off, and fluid is evacuated from the shoulder prior to reimplantation of the bursa.. Nothing is added to the bursa prior to reimplantation. There are no reagents. The bursa tissue is purely the minced bursa tissue removed from the patient, and never leaves the sterile field.
  Arms: Experimental group
Procedure: Control Group(Standard of Care) — Prior to all rotator cuff repairs, a subacromial bursectomy is performed with an oscillating shaver so that the rotator cuff can be visualized and repaired.The current standard of care procedure is to discard this tissue, and then proceed with the rotator cuff repair
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate clinical outcomes, structural integrity, and tendon organization after rotator cuff repair with and without subacromial bursa implantation and to further co-existing research studies performed at The University Of Texas Health Science Center of Houston (UT Health) on Ultrashort Time to Echo-Magnetic Imaging Resonance(UTE-MRI) techniques and their implication for rotator cuff analysis.

ELIGIBILITY:
Inclusion Criteria:

* Present with rotator cuff tears requiring arthroscopic repair as confirmed by a medical expert
* Are able to provide informed consent
* Can commit to study follow-up visits or procedures

Exclusion Criteria:

* Are unable to provide informed consent
* Have additional ipsilateral shoulder complications that will inhibit standard of care treatment and rehabilitation
* Have active infection at operative site
* Have active systemic infection
* Chronic inflammatory condition such as rheumatoid arthritis or lupus
* Has had a corticosteroid injection to the affected shoulder within the six weeks prior to surgery
* Have had prior surgical interventions in the past that have modified the existing natural anatomical arrangement of the rotator cuff/shoulder.
* Non-English speaker

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Change in range of motion | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  range of motion will be measured using a goniometer
Change in strength of shoulder | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  shoulder strength will be measured using handheld dynamometer
Change in pain of shoulder as measured by the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  This is scored form 0-100,lower score means worse pain
Change in functional limitations of shoulder as measured by the Simple Shoulder Test(SST) | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  The SST consists of 12 questions with dichotomous (yes/ no) response options. For each question, the patients indicate that they are able or are not able to do the activity. The scores range from 0 (worst) to 12(best)
Change in pain as assessed by the Visual Analog Scale (VAS) | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  The VAS is scored form 0-10, 0 being no pain and 10 being worst pain
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Computer Adaptive Tests (CATs) | 2 weeks after surgery,6 weeks after surgery,3 months after surgery,6 months after surgery,1 year after surgery,2 years after surgery
  PROMIS CAT-PF is scored on a scale from 20-80, where a higher number indicates higher function

SECONDARY OUTCOMES:
Number of participants with improvement in structural integrity as assessed by postoperative MRI | 6 months post surgery
Number of participants with improvement in structural integrity as assessed by postoperative MRI | 12 months post surgery
Number of participants with improvement in tendon organization as assessed using quantitative postoperative ultrashort magnetic resonance imaging (UTE-MRI) using the same MRI scans from the 6- and 12-month time points. | 6 months post surgery
Number of participants with improvement in tendon organization as assessed using quantitative postoperative ultrashort magnetic resonance imaging (UTE-MRI) using the same MRI scans from the 6- and 12-month time points. | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: James M Gregory, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregory JM, Smith AZ, Zandiyeh P. Effect of Subacromial Bursa Augmentation on Self-Reported and Magnetic Resonance Imaging Outcomes in Arthroscopic Rotator Cuff Repair: A Prospective, Blinded Randomized Clinical Trial. Am J Sports Med. 2026 Jan 18:3635465251407328. doi: 10.1177/03635465251407328. Online ahead of print. PMID 41549447